CLINICAL TRIAL: NCT04902729
Title: Oxytocin Vs Carbetocin at Cesarean Delivery in Women With Morbid Obesity: Double-blind, Randomised Control, Non-inferiority Trial
Brief Title: Oxytocin vs Carbetocin at Cesarean Delivery in Women With Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-03
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Post Partum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; cesarean delivery; carbetocin; duratocin; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin 1IU (Active Comparator): Oxytocin 1IU, administered intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby, followed by infusion 80 mU/min (40 IU in 1L given at a rate of 120 mL/h).
  Interventions: Drug: Oxytocin
- Carbetocin 80mcg (Active Comparator): Carbetocin 80mcg, administered intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Patient is given carbetocin (80mcg) intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Other Names: Duratocin
  Arms: Carbetocin 80mcg
Drug: Oxytocin — Patient is given oxytocin (1IU) intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby, followed by infusion 80 mU/min (40 IU in 1L given at a rate of 120 mL/h).
  Other Names: Pitocin
  Arms: Oxytocin 1IU

SUMMARY:
Postpartum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most commonly used uterotonic drug for the active management of third stage labor, to reduce the risk of PPH and help deliver the placenta. Carbetocin is currently recommended by the SOGC (Society of Obstetricans & Gynecologists of Canada), and is a relatively newer drug with a longer duration of action. It has been previously demonstrated that women with elevated BMI require higher doses of these drugs to induce adequate uterine contraction and dose finding studies undertaken at Mount Sinai Hospital have shown that the ED 90 in obese patients to be carbetocin 80 mcg and oxytocin 1IU. Furthermore, previous studies have indicated that the use of carbetocin over oxytocin in non-obese popultion is associated with reduced bleeding and requirement of additional uterotonic medications. No study has directly compared the two drugs in obese parturients in a head to head clinical trial; therefore a double-blind randomized controlled trial is necessary to show the non-inferiority of carbetocin against the current standard of care at Mount Sinai hospital, which is oxytocin.

DETAILED DESCRIPTION:
Obesity in pregnancy is defined as a Body Mass Index (BMI) above 30 kg/m2 and is often cited as a risk factor for PPH after cesarean delivery.

The World Health organization (WHO) recommends that uterotonic medications are routinely administered at cesarean delivery for the active management of the third stage of labor, both to facilitate delivery of the placenta and to reduce the risk of PPH. The optimal regimen for active management of third stage of labor is yet to be fully determined and obesity adds another layer of complexity and risk, with higher doses required to induce adequate uterine contraction. While oxytocin is the most commonly used drug world-wide, multiple agents are available and there is no clear consensus as to which drug should be first choice. Multiple studies have shown that carbetocin is associated with reduced post-partum bleeding, need for blood transfusion and additional uterotonic medications, in the non-obese population.

The results of this study will provide evidence on the non-inferiority of carbetocin when compared directly to the current standard of care at Mount Sinai hospital, which is oxytocin.

The investigators hypothesize that when administered in equipotent doses, carbetocin would be non-inferior to oxytocin in women with BMI ≥40 kg/m2 undergoing elective cesarean delivery.

The investigators hope to prove that the difference between uterine tone elicited by carbetocin falls within the inferiority margin of -1.2 using a verbal numerical rating score.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥40 kg/m2
* Elective cesarean delivery under spinal, epidural, or combined spinal-epidural anaesthesia
* Written informed consent
* Full term pregnancy (37+0 to 40+6 weeks gestation)
* Non-labouring patients

Exclusion Criteria:

* Refusal to give written informed consent
* Allergy or hypersensitivity to carbetocin or oxytocin
* Laboring patients
* Need for general anaesthesia
* Conditions that predispose to uterine atony and postpartum haemorrhage including but not limited to:
* Placenta previa
* Multiple gestations
* Preeclampsia
* Eclampsia
* Polyhydramnios
* Uterine fibroids
* Previous history of uterine atony and postpartum bleeding
* Bleeding diathesis
* Hepatic, renal, and cardiovascular disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Uterine Tone 3 minutes | 3 minutes
  The primary outcome will be the intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 3 minutes, from the completion of delivery of the drug, utilising a VNRS scale of 0-10.

SECONDARY OUTCOMES:
Uterine Tone 5 minutes | 5 min
  Intensity of uterine tone on a VNRS scale of 0-10 as evaluated by the obstetrician at 5 minutes after completion of injection of the bolus study drug.
Uterine Tone 10 minutes | 10 min
  Intensity of uterine tone on a VNRS scale of 0-10 as evaluated by the obstetrician at 10 minutes after completion of injection of the bolus study drug.
Additional uterotonics - operating room | 1-2 hours, length of surgery will vary
  The use of additional uterotonic agents in the operating room
Additional uterotonics - Post Anesthesia Care Unit (PACU) | 4 hours
  The use of additional uterotonic agents at any time after admission to the recovery area (Post Anesthesia Care Unit (PACU)) until transfer to the post partum ward.
Additional uterotonics - 24 hours | 24 hours
  The use of additional uterotonic agents at any time after discharge from the recovery area (Post Anesthesia Care Unit (PACU)) and up to 24 hours post delivery
Estimated blood loss calculated | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 24 hours after the cesarean section.
Estimated blood loss, visual estimate provided by the obstetrician | 2 hours
  Blood loss in ml, as reported by the obstetrician at the end of the surgery.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Hypertension: systolic blood pressure greater than 120% of baseline | 2 hours
  Systolic blood pressure > 120% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient
Presence of flushing: questionnaire | 2 hours
  Any presence of flushing, from drug administration until end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner W, Boonstra L, Maxwell C, Downey K, Balki M. Oxytocin versus carbetocin at elective Cesarean delivery in parturients with class III obesity: a double-blind randomized controlled noninferiority trial. Can J Anaesth. 2025 Mar;72(3):426-435. doi: 10.1007/s12630-024-02891-2. Epub 2025 Jan 6. PMID 39760981